CLINICAL TRIAL: NCT01269047
Title: Exenatide (Byetta) Vs Pramlintide (Symlin): Role in Post-prandial Hyperglycemia
Brief Title: Use of Exenatide and Pramlintide to Decrease Post-prandial Hyperglycemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rubina Heptulla, Division Chief of Pediatric Endocrinology & Diabetes, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010 -436; R01DK077166 (NIH); NCT00923715 (obsolete NCT alias)
Record Dates: First submitted 2010-12-29; First posted 2011-01-04 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; Symlin; Byetta; CGMS iPro
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide; Exenatide; Insulin; Insulin Aspart; Insulin Lispro; Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pramlintide + Insulin Group (Experimental): These kids will get Pramlintide (Symlin) along with insulin before breakfast and supper.
  Interventions: Drug: Pramlintide
- Exenatide + Insulin Group (Experimental): This group will get Exenatide(Byetta) along with insulin before breakfast and supper.
  Interventions: Drug: Exenatide
- Insulin monotherapy (Active Comparator): This group will be on their regular insulin therapy.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Pramlintide — Start at 15 mcg capped at 60 mcg before breakfast and supper subcutaneously for 4 months
  Other Names: Symlin
  Arms: Pramlintide + Insulin Group
Drug: Exenatide — Start at 1.25 mcg, capped at 5 mcg, subcutaneously, before breakfast and supper for 4 months
  Other Names: Byetta; Type 1 diabetes
  Arms: Exenatide + Insulin Group
Drug: Insulin — Rapid acting and long acting, subcutaneously, according to their regimen for the entire duration of the study.
  Other Names: Novolog; Humalog; Levemir; Lantus
  Arms: Insulin monotherapy

SUMMARY:
The main purpose of the study is to determine the effects of 16 weeks of adjunctive pramlintide or exenatide use on glycemic control in Type 1 Diabetes.

DETAILED DESCRIPTION:
After signing an informed consent, prior to study enrollment, a screening evaluation will be performed in the Clinical Research Center (CRC).

The evaluation will consist of: a medical history, a physical examination with vital signs, Tanner staging, and a waist circumference. The following laboratory tests will be done: CBC, HbA1c, creatinine,Liver function tests, amylase, lipid profile, lipase, urine for pregnancy test (when appropriate) and microalbumin. A urine pregnancy test will be done at each study visit in menstruating females. Also an anti-GAD,IA12, and anti-insulin antibody test will be done, if they were not previously done or if records are not available. Each subject will have a continuous glucose monitoring sensor (CGMS) inserted and will need to wear it for 3 days (72 hours). A person,trained to insert the subcutaneous sensor, will insert the sensor. The sensor is inserted subcutaneously with an injector device. This site insertion is very similar to an insulin pump site insertion. A recorder is attached to the sensor and records blood glucose data for 72 hours. The subject will need to test their blood glucose at least 4 times a day while wearing the sensor. The subject will be asked to keep a log on diet, insulin and exercise while wearing the CGMS. At the end of the 3 day sensing period, the subject will remove the sensor and place the recorder on a charger. The sensor will be brought back by the subject to Visit #1. A Mixed Meal Tolerance Test will be performed at this visit (as described below): Preparation for Mixed Meal Tolerance Test (MMTT)

1. The test will be performed in the morning (between 7 and 10 AM)
2. Test will be conducted only if fasting value by capillary blood glucose meter is between 70-200 mg/dl (3.9-11.1mMol). If the blood glucose prior to start of MMTT is greater than 350 mg/dl, then urine ketones will be measured. If a subject's blood glucose is less than 70 mg/dl before the Mixed Meal Tolerance Test, they will receive 5-10 grams of dextrose 50% by IV. If a subject develops hyperglycemia after the MMTT (which is expected), they will receive a supplemental bolus of fast acting insulin based on their usual insulin sensitivity factor. The subject will be instructed by the study staff on the amount needed. The subject will administer the bolus by themselves
3. Participants on injections will not withhold taking long acting insulin on the morning of the test. Participants can take very short acting insulin (e.g. Humalog or Novolog) up to 2 hours before the test if necessary and then that will be withheld during the test.
4. Participants on insulin pumps will continue with the normal basal rate. Participants can take very short acting insulin (e.g. Humalog or NovoLog) up to two hours before the test if necessary.
5. The participant will be fasting for at least 8 hours and will have had no food or drink (with the exception of water).
6. Local anesthetics may be used as needed to start the I.V. line. Conducting the Mixed Meal Tolerance Test (MMTT)

1. Baseline blood samples will be drawn at -30 minutes; -10 minutes and 0 minutes (immediately before the participant starts drinking the liquid meal) Baseline samples will include glucose, insulin, C-peptide, amylin, GLP-1, glucagon and active ghrelin.

2. The participant will have a standardized liquid meal: Boost HP 6 ml/kg, with a maximum of 360 ml, to be ingested within 5 minutes.

3. Blood samples will be drawn at times: 15, 30, 60, 90 and 120 minutes for glucose, insulin, C-peptide, amylin, GLP-1,active ghrelin and glucagon after the start of ingestion of Boost.

4. After the test is completed, the participant will receive their usual morning dose of short acting insulin analog. The short acting analog will be dosed according to the subject's usual sensitivity factor and insulin to carbohydrate ratio for breakfast as prescribed by the investigator. Subjects on insulin pump therapy will receive a short acting analog via the pump, dosed according to the subject's usual sensitivity factor and insulin to carbohydrate ratio for breakfast as prescribed by the investigator. Subjects will receive a meal tray once the premeal insulin is administered. A total of 107.6 ml of blood will be drawn at the screening visit.

Visit 1 (0 months):

If subjects qualify after screening, they will have the opportunity to enroll in the study. They will meet with a study coordinator in the CRC to make adjustments to their insulin dosage (if necessary) to optimize treatment and improve glycemic control. As shown in the preliminary data section, insulin glargine (Lantus), a long acting analog, may be used when mixed with short acting insulin analogs so as to decrease the total number of injections. This may also increase compliance to the medication regimen. Parental supervision for medication administration will be advised. Hypoglycemic events and adherence to insulin regimen will be noted. Subjects will have vital signs, waist circumference, HbA1C, Glycomark, and a urine pregnancy test (as appropriate).Dual-emission X-ray absorptiometry (DEXA) body scan will be done on this day to estimate total body fat. Patients will also be asked to bring in food diary kept for 3 days so that it can be analyzed for calories being consumed. During the entire study period, subjects will be assessed using a home blood glucose monitor that will electronically transfer data to PI (Glucomon). Data will be reviewed daily for week 1 and 2, and then once a week for week 3 and 4. Starting at week 5, data will be reviewed once every two weeks for the remainder of the study. Contact will be similar for all subjects. Subjects will receive their Glucomon at this visit. At this visit, subjects will be randomized into one of three possible groups.

Randomization: Subjects will be randomized using a random number table. Group 1: Pramlintide + Insulin Group 2: Exenatide + Insulin Group 3: Insulin monotherapy

Study Medications:

Exenatide dosing: Exenatide will be started at 1.25 mcg as previously determined by us in an earlier study. Exenatide injection will be given subcutaneously twice a day (within 30 minutes after the start of the meal) and will be separate from insulin injections. Exenatide dose will be titrated to 2.5 or 5 mcg (depending on response) to keep 2 hr post-prandial blood glucose concentrations below 200 mg/dl. Initially, premeal bolus insulin dose will be reduced by 30%. Basal insulin dose will not be changed. Insulin dose may be increased if pre-meal blood glucose concentrations are greater than 150 mg/dl or to decrease post-prandial hyperglycemia.

Pramlintide dosing: Based on our preliminary studies, pramlintide will be started at 15 mcg and then titrated up to 30-45 mcg and capped at 60 mcg. This will be based on demonstration of acceptable post-prandial glucose excursions without hypoglycemia. Subjects will receive pramlintide subcutaneously twice a day (within 30 minutes after the start of the meal) and will be separate from insulin injections. Initially, premeal bolus insulin dose will be reduced by 30%.Insulin dose may be increased if pre-meal blood glucose concentrations are greater than 150 mg/dl or to decrease post-prandial hyperglycemia.

At the outset, we will decrease premeal bolus insulin dose by 30% for both groups, but insulin may be increased as necessary once the subjects are better able to tolerate the drugs (personal communications regarding unpublished data with Dr. David Maggs, Amylin pharmaceuticals, on the management of exenatide and/or pramlintide with insulin).

Insulin monotherapy: Subjects randomized to insulin monotherapy will continue on either long-acting and short acting insulin analogs or subcutaneous insulin pump therapy. Insulin dose changes will only be made to optimize therapy.

A total of 5.5 ml of blood will be drawn at the Visit 1.

Visit 2 (1 month):

Subjects will have vital signs, waist circumference, HbA1C, Glycomark, and a urine pregnancy test (as appropriate).

Adherence to insulin/medication regimen and adverse event reporting will be obtained.

A total of 5.5 ml of blood will be drawn at the Visit 2.

Visit 3 (4 months):

Subjects will undergo a medical history, physical examination, vital signs, waist circumference, HbA1C, Glycomark,amylase, lipase, Liver function tests, CBC, creatinine, adiponectin, leptin, C-reactive protein, lipid profile, IL-6, and a urine pregnancy test (as appropriate) . Adherence to insulin/medication regimen and adverse event reporting will be obtained. Quality of Life (QOL) questionnaires will be repeated. Additionally, subjects will come in fasting and undergo a MMTT as described in the Screening visit but if subjects are on pramlintide/ exenatide (Byetta) they will receive that dose prior to the boost administration. DEXA scan will be done on this day to estimate total body fat. Patients will also be asked to bring in food diary kept for 3 days so that it can be analyzed for calories being consumed. Each subject with have a continuous glucose monitoring sensor (CGMS) inserted and will need to wear it for 3 days (72 hours). A person, trained to insert the subcutaneous sensor, will insert the sensor. The subject will receive instruction on completion of logsheets and how to properly remove the sensor. Pramlintide and exenatide will be stopped after the subject removes the sensor which is again 3 days from its insertion. Each family would be given a prepaid envelope to mail back the sensor recorder and the remaining study medication. A total of 104.6 ml of blood will be drawn at the Visit 3. Control subjects during the MMTT will receive pramlintide or exenatide as a one time dose without insulin.

Visit 4 (6-7 months):

This will be a post-study visit. Subjects will undergo a medical history, physical examination, vital signs, waist circumference. This visit will be similar to visit 3 for testing and lab work and pregnancy test (as appropriate). Except that the subject will not have DEXA scan and a Continuos Glucose Monitoring Sensor. If the subject received pramlintide previously as study drug in visit 3 they will receive exenatide as a one time dose with the MMTT. QOL questionnaires will be repeated. Adherence to insulin regimen and adverse event reporting will be obtained. Subjects will return their Glucomon and all the blood glucose log books at this visit. A total of 104.6 ml of blood will be drawn at the Visit 4.

During the entire study period, subjects will be assessed using data collected from a study issued home blood glucose monitor. The subject's blood glucose data will be electronically transmitted to the PI ensuring data security and patient privacy. Data will be reviewed daily for weeks 1 and 2, and then once a week for weeks 3 and 4. Starting at week 5,data will be reviewed once every two weeks for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 12 to 21 years.
2. HbA1C less than 9%
3. Subjects must be on intensive insulin management
4. Tanner stage greater than or equal to 3
5. Having Type 1 Diabetes for at least one year
6. Type 1Diabetes defined by ADA criteria and having at least one of the following antibodies a. Anti-GAD (glutamic acid decarboxylase) b. Anti-islet cell 512 (ICA512) c. Anti-insulin
7. Willing to give consent.

Exclusion Criteria:

1. Type 2 diabetes.
2. Having any other chronic condition except hypothyroidism stable on medications.
3. On chronic medications that may affect glucose excursions.
4. Anemia as defined as Hb less than 9 gm/dl.
5. Abnormal amylase, lipase or creatinine (twice normal).
6. Abnormal Liver function tests(three times above normal)
7. Unsupportive family environment as determined by clinicians and/or social workers.
8. Pregnant or lactating mothers

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2009-08; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine West Campus Clinical Research Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 participants were screened. Recruitment began at Baylor College of Medicine, TX in August of 2009 and the last study visit was in July of 2012 at Montefiore Medical Center, Bronx, NY
Period: Overall Study
Arm/Group | Pramlintide + Insulin Group | Exenatide + Insulin Group | Insulin Monotherapy
Started | 13 | 13 | 11
Completed | 12 | 11 | 10
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pramlintide + Insulin Group | Exenatide + Insulin Group | Insulin Monotherapy | Total
Number analyzed (Participants) | 12 | 11 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.0 (3.4) | 15.0 (1.7) | 15.2 (2.1) | 15.7 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 4 | 15
  Male | 5 | 7 | 6 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 8 | 6 | 23
  African American (AA) | 1 | 1 | 1 | 3
  Hispanic | 2 | 2 | 2 | 6
  Mixed (White/AA) | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Post-prandial Blood Glucose Concentration in Both Pramlintide and Exenatide Treated Groups in Acute and Chronic Setting, Compared to Insulin Monotherapy in Type 1 Diabetes Mellitus.
Description: We measured post-prandial blood sugars in both pramlintide and exenatide treated groups in acute and chronic setting, when compared to insulin monotherapy in subjects with Type 1 Diabetes Mellitus
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Acute Pramlintide + Insulin Group: The kids in Exenatide group will get a single dose of Pramlintide at the end of 4 months as part of the 4 hour MMTT.
  The dose of pramlintide used for acute treatment is either 30 mcg or 60 mcg
- Acute Exenatide + Insulin Group: The kids in Pramlintide group will get a single dose of Exenatide at the end of 4 months as part of the 4 hour MMTT.
  The dose of pramlintide used for acute treatment is either 1.25 mcg or 2.5 mcg
- Chronic Pramlintide + Insulin Group: These kids will get Pramlintide (Symlin) along with insulin before breakfast and supper.
  Pramlintide: Start at 15 mcg capped at 60 mcg before breakfast and supper subcutaneously for 4 months
- Chronic Exenatide + Insulin Group: This group will get Exenatide(Byetta) along with insulin before breakfast and supper.
  Exenatide: Start at 1.25 mcg, capped at 5 mcg, subcutaneously, before breakfast and supper for 4 months
- Insulin Monotherapy: These kids received insulin only treatment
Arm/Group | Acute Pramlintide + Insulin Group | Acute Exenatide + Insulin Group | Chronic Pramlintide + Insulin Group | Chronic Exenatide + Insulin Group | Insulin Monotherapy
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 10
mmol/L | 9.03 (1.6) | 8.4 (1.3) | 8.0 (2.0) | 10.2 (1.9) | 10.8 (3.8)
Statistical Analysis 1: Comparison: Acute Pramlintide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.04, ANOVA; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.2 to -0.2], Standard Deviation 2.4
Statistical Analysis 2: Comparison: Acute Exenatide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.008, ANOVA; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-5.8 to -1.3], Standard Deviation 2.7
Statistical Analysis 3: Comparison: Chronic Pramlintide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.003, ANOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.4 to -2.0], Standard Deviation 2.6
Statistical Analysis 4: Comparison: Chronic Exenatide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.37, ANOVA; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-2.3 to 0.98], Standard Deviation 2.0

2. Secondary Outcome: Difference in HbA1C Between the Treatment and the Control Groups
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of HbA1C values
Arm/Group | Acute Pramlintide + Insulin Group | Acute Exenatide + Insulin Group | Chronic Pramlintide + Insulin Group | Chronic Exenatide + Insulin Group | Insulin Monotherapy
Number analyzed (Participants) | 12 | 11 | 11 | 11 | 10
percentage of HbA1C values | 0.30 (0.8) | 0.60 (0.1) | 0.23 (0.6) | 0.40 (1.0) | -0.40 (0.9)
Statistical Analysis 1: Comparison: Acute Pramlintide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.2, t-test, 2 sided; Mean Difference (Final Values) = 0.30, 95% CI 2-sided [-0.21 to 0.81], Standard Deviation 0.8
Statistical Analysis 2: Comparison: Acute Exenatide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.48, t-test, 2 sided; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [-0.25 to 0.50], Standard Deviation 0.6
Statistical Analysis 3: Comparison: Chronic Pramlintide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 0.23, 95% CI 2-sided [-0.12 to 0.57], Standard Deviation 0.6
Statistical Analysis 4: Comparison: Chronic Exenatide + Insulin Group vs Insulin Monotherapy; Test type: Other; p = 1.0, t-test, 2 sided; Mean Difference (Final Values) = -0.004, 95% CI 2-sided [-0.62 to 0.61], Standard Deviation 1.0

ADVERSE EVENTS:
Arm/Group | Pramlintide + Insulin Group | Exenatide + Insulin Group | Insulin Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 1/13 | 1/13 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pramlintide + Insulin Group (N=13) | Exenatide + Insulin Group (N=13) | Insulin Monotherapy (N=11)
Diabetic Ketoacidosis (DKA) (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) — High blood sugars sometimes tend to cause DKA. This could also happen when there is an underlying upper respiratory tract infection or other infections. Symptoms include, nausea, vomitting, abdominal pain etc

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No